CLINICAL TRIAL: NCT03972501
Title: A Single-center, Vehicle-controlled, Study to Evaluate the Safety, Tolerability, and Pharmacodynamics of AZR-MD-001 as Adjunctive Therapy to Conventional Therapeutic Treatment for Meibomian Gland Dysfunction (MGD) or Contact Lens Discomfort (CLD)
Brief Title: An Evaluation of AZR-MD-001 as Treatment for Meibomian Gland Dysfunction (MGD) or Contact Lens Discomfort (CLD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Azura Ophthalmics (Industry)
Collaborators: The University of New South Wales (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SOVS2019-070
Record Dates: First submitted 2019-05-29; First posted 2019-06-03 (Actual); Results first posted 2023-01-25 (Actual); Last update posted 2023-01-25 (Actual); Status verified 2020-03

CONDITIONS: Meibomian Gland Dysfunction (MGD); Contact Lens Discomfort (CLD)
MeSH Terms: conditions — Meibomian Gland Dysfunction

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AZR-MD-001 Vehicle (Placebo Comparator): AZR-MD-001 Vehicle will be dosed up to once daily.
  Interventions: Drug: AZR-MD-001 Vehicle
- AZR-MD-001 Active Dose (Experimental): AZR-MD-001 Active Dose will be dosed up to once daily.
  Interventions: Drug: AZR-MD-001 Active Dose

INTERVENTIONS:
Drug: AZR-MD-001 Vehicle — AZR-MD-001 is an ophthalmic ointment
  Arms: AZR-MD-001 Vehicle
Drug: AZR-MD-001 Active Dose — AZR-MD-001 is an ophthalmic ointment
  Arms: AZR-MD-001 Active Dose

SUMMARY:
SOVS2019-070 is a single-center study of AZR-MD-001 ointment and AZR-MD-001 vehicle in patients with Meibomian Gland Dysfunction (MGD) or Contact Lens Discomfort (CLD).

DETAILED DESCRIPTION:
SOVS2019-070 is a single-center, single-masked (the individual(s) performing efficacy measures will be masked to treatment assignment for the patient(s) they are assessing), vehicle-controlled, randomized, parallel group study of AZR-MD-001 ointment and AZR-MD-001 vehicle in patients with Meibomian Gland Dysfunction (MGD) or Contact Lens Discomfort (CLD).

ELIGIBILITY:
Inclusion Criteria:

* MGD Patients:

  * Evidence of meibomian gland obstruction (based on a meibomian gland secretion (MGS) score of ≤12 for 15 glands of the lower lid) in both eyes at the baseline visit
  * Reported dry eye signs and symptoms within the past 3 months
  * TBUT < 10 seconds in both eyes
* CLD Patients:

  * Evidence of meibomian gland obstruction (based on a meibomian gland secretion (MGS) score of ≤12 for 15 glands of the lower lid) in both eyes at the baseline visit
  * A history of wearing soft contact lenses for at least 6 months
  * Wearing of the soft contact lenses for at least 3 weeks before the baseline visit and wore or attempted to wear lenses at least 4 times a week before the baseline visit.
  * Symptomatic as defined by an answer of "No" at baseline to the question, "Are you able to comfortably wear your lenses as long as you want?"
  * Self-reported history of contact lens dryness/intolerance in the 6 months preceding the baseline visit.
  * Baseline CLDEQ-8 score >12
  * Contact lens may be use during the study as long as they are removed 15 minutes before dosing and not reinserted until at least 15 minutes after dosing.

Exclusion Criteria:

* Uncontrolled ocular disease (except for MGD or CLD) or uncontrolled systemic disease
* Patient has glaucoma or ocular hypertension
* Corneal abnormality or disorder that impacts normal spreading of the tear film or corneal integrity
* BCVA worse than 20/40 in either eye at the baseline visit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2019-10-04 (Actual); Primary Completion 2020-12-11 (Actual); Study Completion 2020-12-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- School of Optometry and Vision Science, University of New South Wales, Sydney, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | AZR-MD-001 Vehicle | AZR-MD-001 Active Dose
Started | 9 (7 patients subsequently completed the Screening period.) | 17 (13 patients subsequently completed the Screening period.)
Completed | 7 | 7
Not Completed | 2 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AZR-MD-001 Vehicle | AZR-MD-001 Active Dose | Total
Number analyzed (Participants) | 9 | 17 | 26
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.8 (19.2) | 21.4 (32.8) | 32.1 (14.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 14 | 19
  Male | 4 | 3 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 6 | 11 | 17
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 6 | 9
Region of Enrollment [Number; unit: participants]
  Australia | 9 | 17 | 26

OUTCOME MEASURES:

1. Primary Outcome: Primary Efficacy for MGD: Change From Baseline to Month 4 in Meibum Gland Secretion Score (MGS).
Description: The MGS can range from 0 (highly abnormal) to 45 (Normal). Meibomian gland assessment was completed using a handheld instrument, Meibomian Gland Evaluator, along the eyelid margin to ensure measurement consistency. A total of 15 glands were evaluated along the lower eyelid margin, consisting of 5 glands located in each of the temporal, central and nasal regions. For each of the 15 glands, expressed secretion characteristics were graded on a 0-3 scale using the methods published by Lane and colleagues (2012).
  Lane SS, DuBiner HB, Epstein RJ, et al. A new system, the LipiFlow, for the treatment of meibomian gland dysfunction (MGD). Cornea. 2012; 31(4): 396-404.
Time Frame: Month 4
Population: Modified Intent to Treat
Measure: Mean (Standard Deviation); unit: Units on the Meibomian Gland Score scale
Arm/Group | AZR-MD-001 Vehicle | AZR-MD-001 Active Dose
Number analyzed (Participants) | 7 | 7
Units on the Meibomian Gland Score scale | 12.1 (10.7) | 16 (11.3)

2. Primary Outcome: Primary Efficacy for MGD: Change From Baseline to Month 4 in Meibomian Glands Yielding Liquid Secretion (MGYLS).
Description: The MGYLS can range from 0 (highly abnormal) to 15 (Normal). Meibomian gland assessment was completed using a handheld instrument, Meibomian Gland Evaluator, along the eyelid margin to ensure measurement consistency. A total of 15 glands were evaluated along the lower eyelid margin, consisting of 5 glands located in each of the temporal, central and nasal regions. The number of glands secreting any liquid were counted using the methods published by Lane and colleagues (2012).
  Lane SS, DuBiner HB, Epstein RJ, et al. A new system, the LipiFlow, for the treatment of meibomian gland dysfunction (MGD). Cornea. 2012; 31(4): 396-404.
Time Frame: Month 4
Population: Modified Intent to Treat
Measure: Mean (Standard Deviation); unit: Units on the MGYLS scale
Arm/Group | AZR-MD-001 Vehicle | AZR-MD-001 Active Dose
Number analyzed (Participants) | 7 | 7
Units on the MGYLS scale | 3.9 (3.2) | 4.1 (4.4)

ADVERSE EVENTS:
Time Frame: 4 Months
Arm/Group | AZR-MD-001 Vehicle | AZR-MD-001 Active Dose
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/13
Other Adverse Events (participants affected / at risk) | 0/7 | 3/13
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AZR-MD-001 Vehicle (N=7) | AZR-MD-001 Active Dose (N=13)
Eye Irritation (Eye disorders) | 0 (0) | 2 (2)
Eye Pain (Eye disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-02-17): https://cdn.clinicaltrials.gov/large-docs/01/NCT03972501/Prot_SAP_000.pdf